CLINICAL TRIAL: NCT00171899
Title: Study Comparing Standard Dose and High-dose Imatinib Mesylate in Patients With Chronic Phase Ph+ CML
Brief Title: Study Comparing Standard Dose and High-dose Imatinib Mesylate in Patients With Chronic Phase Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia (CML)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571ACA09
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic Myelogenous Leukemia; Complete cytogenetic response; Imatinib mesylate; Major molecular response; Chronic phase Ph+ Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

ARMS (1):
- STI571 (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
The study will assess the role of high-dose imatinib mesylate, in patients who have taken imatinib mesylate for at least 1 year at the standard dose, in achieving a major molecular response (a measure of the level of chronic myelogenous leukemia) versus the standard dose.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myelogenous leukemia with Philadelphia chromosome
* 18 years and older
* Patients must have been taking imatinib mesylate standard dose for at least 12 months and have achieved a complete cytogenetic response but not a major molecular response.

Exclusion Criteria:

* Patients with cardiac problems such as congestive heart failure, or myocardial infarction within the last 6 months
* Patients with an uncontrolled medical disease such as uncontrolled diabetes, chronic renal (kidney) disease or active uncontrolled infection.
* Patients with other current primary malignancy or malignancy requiring active intervention

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percent of patients achieving major molecular response at baseline and at last visit

SECONDARY OUTCOMES:
Complete cytogenetic response at baseline and at last visit
Overall survival
Disease progression-free survival
Quality of Life assessment at baseline, last visit
Safety: adverse events and lab parameters, vital signs, physical exam, electrocardiogram, concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Toronto, Canada